CLINICAL TRIAL: NCT04985045
Title: Determination of Menstrual Health and Genital Hygiene Status in Women With Cerebral Palsy
Brief Title: Menstrual Health and Genital Hygiene Status in Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Özge Çoban (Other)
Responsible Party: Sponsor-Investigator, Özge Çoban, Universith of Health Science, Health Science Faculty, Lecturer, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Other Study IDs: 2021/191
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Menstrual Problem; Cerebral Palsy; Women's Health
MeSH Terms: conditions — Menstruation Disturbances; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Healthy women will be included
  Interventions: Other: Evaluation
- Cerebral palsy group: Women with cerebral palsy will be included
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Individuals' menstrual status, pain, menstrual symptoms and genital hygiene behaviors will be evaluated.

SUMMARY:
There is little information about the menstrual health and genital hygiene behaviors of young women with CP. The most important reason for this is that women with CP did not meet the inclusion criteria and were excluded from the study. This may lead to a knowledge gap that limits the design of approaches that can help women and families with CP. Therefore, this study was planned to determine menstrual health and genital hygiene behaviors in women with CP.

ELIGIBILITY:
Inclusion Criteria:

for women with cerebral palsy (CP)

1. Participating in the research voluntarily,
2. Being diagnosed with CP
3. To be GMFCS level I-II-II
4. to be 10-30 years old,
5. Being able to read and write Turkish,
6. Not having any mental problems that prevent cooperation and understanding,
7. Being a woman
8. To have menstruated at least once.

For healthy women

1. Participating in the research voluntarily,
2. to be 10-30 years old,
3. Being able to read and write Turkish,
4. Not having any mental problems that prevent cooperation and understanding,
5. Being a woman
6. To have menstruated at least once.

Exclusion Criteria:

1. Having a history of pregnancy
2. Having an acute genital infection
3. To have undergone gynecological surgery.

Ages: 10 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Women with menstrual cycle
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual Pain | A month
  The highest pain intensity experienced by individuals during the menstrual period will be determined using the visual analog scale. Individuals will be asked to determine the highest pain intensity experienced during menstruation on a straight line from 0 to 10 cm. In this chart, "0" means I have no pain, "10" means I have unbearable pain. Facial expressions will be added below the line to increase the clarity of the assessment. At the same time, adolescents will be asked to mark where the pain is on the front and back body images.
Menstruation-related symptoms | A month
  Menstruation-related symptoms of individuals will be determined using the "Menstruation Symptom Scale (MSS)". The Menstruation Symptom Scale was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. It is a widely used scale in studies conducted in many different countries. The scale consists of 22 items questioning the symptoms related to menstruation and is scored in a five-point Likert type as never (1), rarely (2), sometimes (3) often (4) and always (5). The total score of MSS is calculated by taking the mean score of all items in the scale. An increase in the total score indicates an increase in the severity of menstrual symptoms. The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints', 'Menstrual Pain' and 'Coping Methods'.
Genital Hygiene status | A month
  The genital hygiene behaviors of individuals will be evaluated using the "Genital Hygiene Behaviors Scale (GHDS)". The GHQ scale is a five-point Likert-type scale consisting of 23 items and 3 sub-dimensions developed by Karahan (2017). The level of agreement with the statements is scored as "Totally agree (5)", Agree (4), Undecided (3) Disagree (2), Completely disagree (1). The total score is obtained by adding the point values of the answers given to all the statements. The first 12 items of the scale include general hygiene habits, 13-20. substances, menstrual hygiene, 21-23. items are intended to determine abnormal finding awareness. 5 items of the scale have reverse entries. The total score varies between 23-115. Higher scores indicate improved genital hygiene.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turker D, Dogan H, Coban O, Goksuluk MB, Ozengin N, Un Yildirim N. Menstrual health and genital hygiene status in adolescent girls and young women with cerebral palsy. Women Health. 2023 Apr;63(4):243-250. doi: 10.1080/03630242.2023.2171175. Epub 2023 Feb 12. PMID 36775296